CLINICAL TRIAL: NCT07074080
Title: Comparative Study of Hand vs. Foot Chest Compressions in a Simulated Environment: Assessment of Compression Effectiveness and Rescuer Fatigue
Brief Title: Hand vs. Foot Chest Compressions in Simulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FOOT-CPR 2025
Record Dates: First submitted 2025-06-05; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Arrest (CA)
Keywords: CA (Cardiac Arrest); CPR (Cardiopulmonary Resuscitation); CPR-FOOT (Foot-based Cardiopulmonary Resuscitation); (HRV) Heart Rate Variability
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: This is a single-center, randomized, crossover, and controlled study conducted at the Skills Laboratory of the Faculty of Medicine and Health Sciences, Campus Clínic. Each participant will serve as their own control, performing chest compressions using both the hands and the foot. The order of the compression method (manual or foot) will be randomly assigned, with participants subsequently performing the alternative method they did not initially complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HM - Hand Method (Active Comparator)
  Interventions: Other: Performance of standard chest compressions with the upper limbs.
- FM - Foot Method (Experimental)
  Interventions: Other: Performing chest compressions on a mannequin using the foot

INTERVENTIONS:
Other: Performing chest compressions on a mannequin using the foot — Performing chest compressions on a mannequin using the foot
  Arms: FM - Foot Method
Other: Performance of standard chest compressions with the upper limbs. — Performance of standard chest compressions with the upper limbs.
  Arms: HM - Hand Method

SUMMARY:
Cardiopulmonary resuscitation (CPR) is essential in the management of cardiorespiratory arrest (CA) to improve survival rates. High-quality chest compressions are the primary intervention to maintain circulation and oxygenation of vital organs during cardiac arrest, making them a key determinant in CPR effectiveness.

Guidelines emphasize that the quality of chest compressions is a critical factor in the effectiveness of basic life support (BLS). To ensure efficacy, a compression rate of 100 to 120 per minute is recommended, with a depth of at least 5 cm but not exceeding 6 cm, proper arm and hand alignment, full chest recoil after each compression, minimal interruptions during CPR, and rescuer rotation every 2 minutes to prevent performance decline due to fatigue.

As we can see, these guidelines refer to performing compressions using the upper limbs. However, it is essential to acknowledge that some individuals have physical limitations that may impair their ability to apply effective force with their upper limbs (e.g., amputations, fractures, neuromuscular dysfunctions). This presents important challenges regarding accessibility and inclusive CPR training. In addition, the use of the lower extremities has been proposed as an alternative to potentially reduce rescuer fatigue, although evidence regarding its effectiveness and impact on physiological fatigue is still limited.

There are studies comparing chest compressions performed with the hands (Hands Method, HMM) and with the feet (Foot Method, FMM); however, these studies have certain limitations and a limited number of participants. Although the quality of CPR was lower when using the feet technique, the results were positive.

However, to date, no specific guidelines have been established on how to perform CPR using the feet (Foot CPR), and it remains unclear whether the position of the feet on the chest or whether compressions are performed with or without shoes are variables that influence compression quality.

Furthermore, during CPR, it is recommended to rotate rescuers every 2 minutes when two or more rescuers are available due to fatigue associated with the procedure. Current evidence suggests that CPR is most effectively performed in the kneeling position, rather than standing or using a stool, due to the lower levels of fatigue in this position.

Traditionally, exercise-induced fatigue is assessed using subjective perception of exertion (RPE), performance monitoring (e.g., power or speed), or biochemical markers (e.g., blood lactate). More recently, heart rate variability (HRV) has been proposed as a valuable tool for assessing the autonomic nervous system response to exercise stress and quantifying physiological fatigue.

After exercise, especially if it is intense or prolonged, the body experiences significant physiological stress. This stress affects multiple systems, including the cardiovascular and autonomic nervous systems. Post-exercise fatigue is a complex sensation involving muscular, metabolic, and neuronal factors. Therefore, HRV becomes a valuable biomarker.

Numerous studies have shown a correlation between decreased HRV and the subjective perception of fatigue after exercise. People with lower heart rate variability (HRV) after exercise tend to report higher levels of fatigue. HRV analysis provides an objective and physiological measure of the stress the body experiences after short-duration, high-intensity exercise, such as that performed during resuscitation.

Therefore, measuring HRV after 2 minutes of chest compressions can indicate the degree of exercise-induced physiological fatigue, which could vary depending on the technique used (Hands-on CPR [H-CPR] vs. Feet-on CPR [F-CPR]).

Efforts to improve outcomes should focus on optimizing the chain of survival through training in Basic Life Support and Automated External Defibrillation (BLS + AED). Offering these courses to the general population presents significant challenges in terms of accessibility and implementation of comprehensive and inclusive training.

The objective of our randomized simulation study using mannequins, with a population of Basic Life Support students, was to compare the quality of chest compressions and the fatigue produced by this technique, in compressions performed with the hands and with the foot.

DETAILED DESCRIPTION:
This is a single-center, randomized, crossover, controlled study conducted in the Skills Laboratory of the Faculty of Medicine and Health Sciences, Campus Clínic. Each participant will act as their own control, performing chest compressions with both hands and their foot. The order of compression method (hand or foot) will be randomly assigned, and participants will subsequently perform the alternative method they did not initially complete.

Participants will be enrolled in a Basic Life Support and Automated External Defibrillation (BLS+AED) course from the Catalan Resuscitation Council - European Resuscitation Council.

Data collection will be consecutive and open-label.

Variable-size block randomization, generated using statistical software, will be used to ensure balanced assignment of participants to the study groups while maintaining unpredictability.

To implement this randomization, the R programming language will be used, widely used in scientific research and statistical analysis due to its robustness and reliability. R offers specialized tools for this type of randomization, ensuring a rigorous, transparent, and reproducible process.

We will use the R package blockrand, specifically designed for efficient and controlled block randomization.

Primary objectives:

To compare the depth of uninterrupted chest compressions (without ventilation) delivered over a 2-minute period during a simulated cardiac arrest on the floor, using either the hands (HM) or feet (FM).

To assess CPR-associated fatigue in the two groups using:

Subjective measures: Rating of perceived exertion (Borg score). Direct objective measures: Use of a wearable health monitoring device (abdominal strap-based) to measure rescuer heart rate variability (HRV), a parameter correlated with fatigue during CPR.

Indirect objective measures: heart rate and oxygen saturation.

Data will be collected using the SkillReporter® app (Laerdal Medical®) during 2 minutes of continuous chest compressions on a Resusci Anne QCPR manikin, a certified medical-grade abdominal strap (Movesense®), and a pulse oximeter.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Signed informed consent
* First-year postgraduate trainees in health-related fields such as medicine or nursing
* Enrolled in a Basic Life Support and Automated External Defibrillation (BLS+AED) course from the Consell Català de Resuscitació - European Resuscitation Council

Exclusion Criteria:

* Physical limitations preventing chest compressions with hands or feet
* Contraindications for physical exercise (e.g., arthritis, heart disease, advanced lung disease, severe physical disability, morbid obesity, chronic fatigue, pregnancy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2025-06-06 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
MEAN CHEST COMPRESSION DEPTH | One day
  Data will be collected using the SkillReporter® application (Laerdal Medical®) during 2 minutes of continuous chest compressions on a Resusci Anne QCPR manikin.
  Primary Variable:
  Mean chest compression depth: To compare the mean depth of uninterrupted chest compressions (without ventilations) performed over a 2-minute period during a simulated cardiac arrest on the floor using the hands (HM) or the feet in both positions (FM-S and FM-T).
DFA α1 (DETRENDED FLUCTUATION ANALYSIS - α1) | One day
  DFA α1 - Short-term scaling exponent from Detrended Fluctuation Analysis (DFA) is a nonlinear HRV metric derived from detrended fluctuation analysis, representing short-term fractal scaling behavior of RR intervals. Assesses fractal-like correlation properties of heart rate time series over short time scales. It provides insights into the complexity and self-regulation of autonomic control. Values closer to 1.0 indicate healthy, adaptable systems, while deviations may suggest altered autonomic regulation.
  Change in heart rate variability (HRV), measured before and after performing the two minutes of CPR using a certified medical-grade abdominal band device (Movesense®).
  HRV is a non-invasive indicator of autonomic nervous system (ANS) activity and is known to be affected by physical fatigue and physiological stress.

SECONDARY OUTCOMES:
OVERALL COMPRESSION SCORE | One day
  Overall compression score (%): A variable created by Laerdal Medical® reflecting how closely CPR performance aligns with ERC Guidelines. Deviations reduce the score from 100%. The score incorporates depth, rate, incomplete release, number of compressions per cycle, and hand/foot positioning.
TOTAL NUMBER OF COMPRESSIONS | One day
  Total number of compressions will be collected using the SkillReporter® application (Laerdal Medical®) during 2 minutes of continuous chest compressions on a Resusci Anne QCPR manikin
COMPRESSION / DESCOMPRESSION RATIO | One day
  This variable refers to the ratio between the duration of the downward chest compression and the upward chest recoil (decompression). Compression/decompression ratio will be collected using the SkillReporter® application (Laerdal Medical®) during 2 minutes of continuous chest compressions on a Resusci Anne QCPR manikin
CORRECT COMPRESSION DEPTH | One day
  Correct compression depth (%): percentage of chest compressions with a depth between 5 and 6 cm. Data will be collected using the SkillReporter® application (Laerdal Medical®) during 2 minutes of continuous chest compressions on a Resusci Anne QCPR manikin
COMPRESSION RELEASE | One day
  Compression release (%) refers to the percentage of chest compressions in which full chest recoil was achieved. Compression release (%) will be collected using the SkillReporter® application (Laerdal Medical®) during 2 minutes of continuous chest compressions on a Resusci Anne QCPR manikin
MEAN COMPRESSION RATE | One day
  Mean compression rate refers to the average number of chest compressions delivered per minute (cpm). Data will be collected using the SkillReporter® application (Laerdal Medical®) during 2 minutes of continuous chest compressions on a Resusci Anne QCPR manikin
CORRECT HANDS/FEET POSITION | One day
  Correct hand/feet position (%): Correct Hand/Feet Position (%) refers to the percentage of chest compressions performed with the hands or feet placed correctly Data will be collected using the SkillReporter® application (Laerdal Medical®) during 2 minutes of continuous chest compressions on a Resusci Anne QCPR manikin
TOTAL NUMBER OF BREAKS | One day
  Total number of breaks: The total count of pauses or interruptions during chest compressions Data will be collected using the SkillReporter® application (Laerdal Medical®) during 2 minutes of continuous chest compressions on a Resusci Anne QCPR manikin
BORG SCALE | One day for each participant (3 weeks in total).
  The Borg Scale measures perceived exertion or subjective intensity of effort during chest compressions. The Borg scale will be used before and after compressions to assess perceived fatigue in all groups.
STANDARD DEVIATION OF NN INTERVALS (SDNN) | One day
  SDNN (Standard Deviation of NN intervals): Reflects overall heart rate variability (HRV) by measuring the standard deviation of all normal-to-normal (NN) intervals. It indicates general autonomic activity and long-term components of variability. Change in heart rate variability (HRV), measured before and after performing the two minutes of CPR using a certified medical-grade abdominal band device (Movesense®).
  HRV is a non-invasive indicator of autonomic nervous system (ANS) activity and is known to be affected by physical fatigue and physiological stress.
ROOT MEAN SQUARE OF SUCCESSIVE DIFFERENCES (RMSSD) | One day
  RMSSD (Root Mean Square of Successive Differences): Represents the short-term heart rate variability (HRV by calculating the square root of the mean squared differences between adjacent NN intervals. It is primarily influenced by parasympathetic (vagal) activity. Change in heart rate variability (HRV), measured before and after performing the two minutes of CPR using a certified medical-grade abdominal band device (Movesense®).
  HRV is a non-invasive indicator of autonomic nervous system (ANS) activity and is known to be affected by physical fatigue and physiological stress.
LOW FREQUENCY (LF) | One day
  Low Frequency (LF) refers to the power of heart rate variability (HRV) within the frequency range of 0.04 to 0.15 Hz in spectral (frequency-domain) analysis.
  This means it reflects oscillations in heart rate that occur every 7 to 25 seconds.Represents a combination of sympathetic and parasympathetic modulation, commonly associated with baroreflex activity.
  Change in heart rate variability (HRV), measured before and after performing the two minutes of CPR using a certified medical-grade abdominal band device (Movesense®).
  HRV is a non-invasive indicator of autonomic nervous system (ANS) activity and is known to be affected by physical fatigue and physiological stress.
HIGH FREQUENCY (HF) | One day
  High Frequency (HF) refers to the power of heart rate variability within the frequency range of 0.15 to 0.40 Hz in spectral (frequency-domain) analysis.
  This corresponds to oscillations in heart rate occurring approximately every 2.5 to 7 seconds, which are strongly linked to respiratory activity. HF (High Frequency, 0.15-0.40 Hz): Reflects parasympathetic activity and is related to respiratory sinus arrhythmia.
  Change in heart rate variability (HRV), measured before and after performing the two minutes of CPR using a certified medical-grade abdominal band device (Movesense®).
  HRV is a non-invasive indicator of autonomic nervous system (ANS) activity and is known to be affected by physical fatigue and physiological stress.
LOW FREQUECY (LF) /HIGH FREQUENCY (HF) RATIO | One day
  The LF/HF ratio is the ratio of Low Frequency (LF) power to High Frequency (HF) power in the spectral analysis of heart rate variability (HRV). LF/HF Ratio Indicates the balance between sympathetic and parasympathetic nervous system activity. An increased ratio may reflect sympathetic dominance.
  Change in heart rate variability (HRV), measured before and after performing the two minutes of CPR using a certified medical-grade abdominal band device (Movesense®).
  HRV is a non-invasive indicator of autonomic nervous system (ANS) activity and is known to be affected by physical fatigue and physiological stress.
JT/RR ratio | One day
  The JT/RR ratio is the ratio between the JT interval and the RR interval on an ECG.
  Change in heart rate variability (HRV), measured before and after performing the two minutes of CPR using a certified medical-grade abdominal band device (Movesense®). HRV is a non-invasive indicator of autonomic nervous system (ANS) activity and is known to be affected by physical fatigue and physiological stress.
SpO₂ | one day
  SpO₂: Oxygen saturation measured by a portable digital pulse oximeter before and after 2 min of chest compressions
PULSE RATE | one day
  Pulse rate: Number of heartbeats per minute (bpm), measured via pulse waveform by a portable digital pulse oximeter before and after 2 minutes of chest compressions.

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Medicina de La Universidad de Barcelona, Barcelona, BARCELONA, Spain

IPD SHARING:
Plan to Share IPD: Yes
At the time of inclusion in the study and after signing the informed consent, personal data will be coded. The data (with coded information) will be collected in an Excel® database, which will be accessible to the collaborating researchers. Access to identifiable data will be restricted to the principal investigator, who will keep it for a maximum of 5 years.